CLINICAL TRIAL: NCT06333535
Title: The Effect of Foot and Abdominal Massage Applied to After Colonoscopy on Abdominal Distention, Pain and Patient Satisfaction
Brief Title: Foot and Abdominal Massage Applied to After Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Turkan Ulker, RN, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/568
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Abdominal Pain; Distention; Satisfaction, Patient
MeSH Terms: conditions — Abdominal Pain; Dilatation, Pathologic; Patient Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Foot massage group (Experimental): Stage 1/Pretest: After the colonoscopy procedure, after the patients regained consciousness in the recovery unit, the Patient Introduction Form, Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were filled out.
  2nd Stage/Intervention: The patients were massaged on both feet in accordance with the foot massage instructions.
  3rd Stage / 30th minute: Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded. .
  4th Stage / 2nd hour: Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded.
  5th Stage / 4th Hour Abdominal Pain NRS Scale Form, Abdominal Distension NRS Scale Form and satisfaction (NRS satisfaction) scores were directed to the patients and recorded.
  Interventions: Other: foot massage
- Abdominal massage group (Experimental): Stage 1/Pretest: After the colonoscopy procedure, after the patients regained consciousness in the recovery unit, the Patient Introduction Form, Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were filled out.
  2nd Stage/Intervention: The patients were massaged in the abdominal area in accordance with the abdominal massage instructions.
  3rd Stage / 30th minute: Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded. .
  4th Stage / 2nd hour: Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded.
  5th Stage / 4th Hour Abdominal Pain NRS Scale Form, Abdominal Distension NRS Scale Form and satisfaction (NRS satisfaction) scores were directed to the patients and recorded.
  Interventions: Other: abdominal massage
- Foot and Abdominal massage group (Experimental): Stage 1/Pretest: After the colonoscopy procedure, after the patients regained consciousness in the recovery unit, the Patient Introduction Form, Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were filled out.
  2nd Stage/Intervention: The patients were massaged in the abdominal area in line with the abdominal massage instructions, and then both feet were massaged in line with the foot massage instructions.
  3rd Stage / 30th minute: Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded.
  4th Stage / 2nd hour: Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded.
  5th Stage / 4th Hour Abdominal Pain NRS Scale Form, Abdominal Distension NRS Scale Form and satisfaction (NRS satisfaction) scores were directed to the patients and recorded.
  Interventions: Other: foot and abdominal massage
- Control group (No Intervention): Stage 1/Pretest: After the colonoscopy procedure, after the patients regained consciousness in the recovery unit, the Patient Introduction Form, Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were filled out.
  Stage 2/Attempt: No attempt was made. 3rd Phase / 30th minute: Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded.
  4th Stage / 2nd hour: Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded.
  5th Stage / 4th Hour Abdominal Pain NRS Scale Form and Abdominal Distension NRS Scale Form were administered to the patients and recorded.

INTERVENTIONS:
Other: foot massage — foot massage
  Arms: Foot massage group
Other: abdominal massage — abdominal massage
  Arms: Abdominal massage group
Other: foot and abdominal massage — foot and abdominal massage
  Arms: Foot and Abdominal massage group

SUMMARY:
The aim of this study was to determine the effect of foot and abdominal massage applied to after colonoscopy on abdominal distention, pain and patient satisfaction.This was a randomized controlled experimental study conducted at the Colonoscopy unit in Medica Faculty Hospital . Participants assigned to the intervention group-1 received foot massages after colonoscopy, participants assigned to the intervention group-2 received abdominal massages after colonoscopy and participants assigned to the intervention group-3 received foot and abdominal massages after colonoscopy. Participants assigned to the control group received only "routine care" after colonoscopy. The abdominal pain, distension and satisfaction levels of the patients evaluated using the Numerical Rating Scale

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of foot and abdominal massage applied to after colonoscopy on abdominal distention, pain and patient satisfaction.This was a randomized controlled experimental study conducted at the Colonoscopy unit in Medica Faculty Hospital . Participants meeting inclusion criteria were assigned to intervention and control groups using a random. Participants assigned to the intervention group-1 received foot massages after colonoscopy, participants assigned to the intervention group-2 received abdominal massages after colonoscopy and participants assigned to the intervention group-3 received foot and abdominal massages after colonoscopy. Participants assigned to the control group received only "routine care" after colonoscopy. The abdominal pain, distension and satisfaction levels of the patients evaluated using the Numerical Rating Scale

ELIGIBILITY:
Inclusion Criteria:

* Being of 18 years of age and above
* Applying for colonoscopy for diagnosis and treatment,
* Being conscious and oriented to place, person and time,
* Having pain after the procedure,
* No communication barriers,
* Able to communicate in Turkish,
* Individuals who gave written consent to participate in the research were included in the study.

Exclusion Criteria:

* Having any psychiatric disease,
* Those who have previously had bowel resection or another bowel surgery,
* Those with colostomy and ileostomy,
* Those with percutaneous endoscopic gastrostomy,
* Those with Inflammatory Bowel Disease,
* Having a history of malignant intestinal obstruction in their health history,
* Diagnosed with colon cancer,
* Those with umbilical/abdominal hernia,
* Having an open wound in the abdominal and/or foot area,
* Those with active lower gastrointestinal system bleeding,
* Those with celiac disease,
* Patients with FMF disease were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
abdominal pain | The end of the colonoscopy (0. Min), the end of intervention 30.min., 2. hour and 4. hour ]
  Abdominal pain evaluated with the Numerical Rating Scale Scale Zero = minimum value Ten = maximum value
Abdominal distension | The end of the colonoscopy (0. Min), the end of intervention 30.min., 2. hour and 4. hour
  Abdominal distension evaluated with the Numerical Rating Scale Scale Zero = minimum value Ten = maximum value
Patient Satisfaction | The end of intervention 4. hour
  Satisfaction evaluated with the Numerical Rating Scale Scale Zero = minimum value Ten = maximum value

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)